CLINICAL TRIAL: NCT01891136
Title: Pilot Study: Oral Peanut Immunotherapy for Peanut Allergic Patients
Brief Title: Oral Peanut Immunotherapy for Peanut Allergic Patients
Acronym: PnOIT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Wesley Burks, MD, Professor of Pediatrics, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-2298; NCT00598039 (obsolete NCT alias)
Record Dates: First submitted 2013-05-24; First posted 2013-07-02 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Peanut Hypersensitivity
Keywords: Peanut allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peanut protein (Experimental): Subjects to receive varying amounts of peanut protein as peanut oral immunotherapy.
  Interventions: Drug: Peanut protein

INTERVENTIONS:
Drug: Peanut protein — Subjects will receive increasing amounts of peanut protein over the modified rush phase and the build-up phase of the protocol. Once the subject reaches the maintenance phase of the study, they will remain on that dose until they reach the oral food challenges at the end of the study.
  Other Names: Peanut OIT

SUMMARY:
This is a study to determine if peanut oral immunotherapy (OIT) would desensitize or tolerize peanut allergic patients to peanuts in order prevent peanut allergic reactions.

DETAILED DESCRIPTION:
The goal of this proposal is to develop peanut OIT for patients with peanut allergic reactions. This approach is designed to utilize our extensive knowledge of the allergens involved in peanut hypersensitivity to devise an immunotherapeutic approach that would lower the risk of anaphylactic reactions and would down regulate peanut-specific T cells in peanut-allergic patients. Previous attempts to utilize peanut-specific immunotherapy (IT) have been unsuccessful primarily because of the side effects of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 1 and 16 years of age
* Diagnosed peanut allergy by either: 1) a positive prick skin test to peanut, CAP FEIA of 15 or greater and a history of significant clinical symptoms within one hour after ingestion of peanuts or 2) a positive prick skin test to peanut, CAP FEIA of ≥ 7 and a history of a clinical reaction to peanut ingestion within the past 6 months.
* A family that will be able to be compliant with all study visits.

Exclusion Criteria:

* Subjects with a history of severe anaphylaxis to peanut
* Subjects with a medical history that would prevent a DBPCFC/OFC to peanut The medical history that would prevent the DBPCFC to peanut would be a prior history of an open peanut challenge in which the patient experienced hypotension which required fluid resuscitation, respiratory compromise which necessitated ventilatory support, or poorly controlled asthma as evidenced by an forced expiratory volume in 1 second (FEV1) < 80% of predicted, or FEV1/FVC (forced vital capacity) < 75%, with or without controller medications
* Subjects unable to cooperate with challenge procedures or unable to be reached by telephone for follow-up
* Pregnant or lactating
* Allergy to oat

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2004-04; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The percentage of peanut-allergic patients achieving clinical desensitization to peanut, assessed after up to five years of OIT. | 2 to 5 years
  Clinical desensitization will be measured with an oral food challenge (OFC) to peanut conducted while on OIT therapy.
Clinical desensitization will be measured with an oral peanut challenge conducted while on OIT therapy. | 2 to 5 years
  Clinical tolerance will be measured with an oral peanut challenge conducted four weeks after discontinuing OIT.

SECONDARY OUTCOMES:
Changes in number of antigen-specific lymphocytes. | 2 to 5 years
  The investigators will examine the role of OIT on peanut-specific T cell responses by enumerating specific T cell subsets, including T regulatory cells, pre- and post-treatment.
Changes in function of antigen-specific lymphocytes. | 2-5 years
  The investigators will examine the role of OIT on peanut-specific T cell responses by analyzing cell signaling, gene expression, and cytokine production, pre- and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States